CLINICAL TRIAL: NCT06566638
Title: Safety, Tolerability and Performance of the NucleoCapture Extracorporeal Therapeutic Apheresis Device in the Reduction of Circulating cfDNA/NETs in Subjects With Pancreatitis
Acronym: NUC-SAP1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Santersus AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHS0096
Record Dates: First submitted 2024-08-07; First posted 2024-08-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-07

CONDITIONS: Acute Pancreatitis; Organ Failure, Multiple
Keywords: Acute pancreatitis; NucleoCapture; Extracorporeal; Apheresis; Neutrophil extracellular traps
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the control arm (SOC) or the treatment arm (SOC plus NucleoCapture) in a 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC plus NucleoCapture (Experimental): Participants in the treatment arm will receive SOC plus three apheresis treatment sessions with the NucleoCapture device. The device consists of 100ml NucleoCapture selective adsorber.
  Interventions: Device: NucleoCapture device
- SOC (No Intervention): Participants in the SOC arm will receive SOC alone, in accordance with ESICM guidelines.

INTERVENTIONS:
Device: NucleoCapture device — 100ml NucleoCapture selective DNA adsorber.
  Arms: SOC plus NucleoCapture

SUMMARY:
This is a single-centre, randomised-controlled, open-label, feasibility study to assess the safety, tolerability and performance of the NucleoCapture extracorporeal apheresis device in the reduction of circulating cell-free DNA (cfDNA)/Neutrophil Extracellular Traps (NETs) in patients with severe acute pancreatitis.

DETAILED DESCRIPTION:
This study investigates the safety, tolerability and performance of the NucleoCapture extracorporeal apheresis device in patients with acute pancreatitis. Acute pancreatitis is one of the leading gastrointestinal disorders that require urgent clinical care and is increasing in incidence.

cfDNA/NET therapeutic apheresis with NucleoCapture is indicated for the treatment of diseases in which excessive levels of cfDNA/NETs are found, such as acute pancreatitis. Participants will be randomised to receive either standard of care (SOC) alone or SOC plus NucleoCapture treatment. SOC will be according to the current guidelines described by the European Society of Intensive Medicine (ESICM). Participants in the SOC plus NucleoCapture arm will receive one treatment session with NucleoCapture per day, for the first three days. Each treatment session with NucleoCapture will last for up 6 hours, aiming to treat 4.5 plasma volumes. Treatment sessions with NucleoCapture treating less than 3.5 plasma volumes will be counted as incomplete and the treatment session will be repeated on the following day, up to day 5 maximum.

Assessments will take place for all participants whilst in the Intensive Care Unit (ICU) on days 1 to 5, 7, 14, 21 and 28, and at 90 days post discharge to ward-based care. Participants transferred to ward-based care before day 28 will receive no further study assessment visits from the point of transfer to ward-based care, apart from day 28 in which participants will receive a final study assessment visit and a patient reported outcome assessment (PROM) 90 days post discharge to ward-based care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 or over
2. Acute pancreatitis (following revised Atlanta definition of 2 out of typical pain, serum amylase >3x normal range and/or CT/MRI imaging consistent with pancreatitis)
3. Any aetiology
4. Acute respiratory (PaO2/FiO2 <300), cardiovascular (systolic BP <90 or any inotropic therapy) or renal failure (serum creatinine >170 µmol/l, or deterioration of >50% eGFR if pre-existing renal disease or urine output <0.5ml/kg/hr for 3 consecutive hours) presenting at any point during the index admission and persistent after 12 h of fluid resuscitation, but for not more than 72 hours
5. Have provided written informed consent or consent is given by the patient's legally designated representative or an independent physician (if possible, according to local law).

   Exclusion Criteria:
6. The use of other non-routine extracorporeal treatments such as very high flux renal replacement therapy (>60ml/kg/h total exchange), use of high cut off filters or other non-routine extracorporeal treatment columns such as Cytosorb, Toramyxcin, etc).
7. Presence of severe multiple organ failure at the point of enrolment as evidenced by:

   * Severe refractory vasoplegic failure

     * Norepinephrine dose > 0.60 μg/kg/min
     * Use of epinephrine
   * Concomitant cardiogenic shock, clinically suspected or cardiac index <2.2 L/min/m2 if measured

     * Use of dobutamine, epinephrine, phosphodiesterase inhibitors or levosimendan
   * Coagulopathy as defined by Platelet count <50x10^9/L
8. Calculated Plasma Volume greater than 5000ml as determined by the following formula:

   Vplasma = Vblood x (1 - haematocrit)

   Where:

   Vplasma = PV Vblood = an estimation of total blood volume (TBV; according to Nadler's formula, incorporating height, weight and sex).

   A TBV calculator is available at https://www.omnicalculator.com/health/blood-volume
9. Known liver cirrhosis (histologically proven or clinically suspected)
10. Active bleeding
11. Known citrate intolerance if citrate is required for therapeutic apheresis
12. Known heparin allergy if heparin is required for therapeutic apheresis
13. Known metastatic disease with life expectancy of <12 months and ECOG score of at least 2
14. Known haematological malignancy if not in remission
15. Known solid organ transplant and concomitant use of immunosuppression
16. Known long term oxygen therapy or Home oxygen use
17. Dialysis dependent Chronic Kidney Disease (CKD Stage 5-D)
18. Planned or impending dialysis
19. Prior use of cardiopulmonary resuscitation (CPR) in current admission
20. Requirement for extracorporeal membrane oxygenation (ECMO)
21. Patient expected to die within 48 hours of admission to ICU
22. Known allergy to components of NucleoCapture (Sepharose beads and linker histone H1.3)
23. Pre-existing disease of the exocrine pancreas including chronic pancreatitis, recurrent acute pancreatitis, pancreatic malignancy and/or history of pancreatic surgery
24. Chronic neuromuscular disease affected breathing
25. Current Participation in another interventional clinical study
26. Pregnancy (as established by the presence of beta human chorionic gonadotropin in urine or blood)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The amount of cfDNA/NETs in the plasma of patients with severe acute pancreatitis after each NucleoCapture treatment. | Within 6 hours from the baseline once 4.5 plasma volumes has been treated.
  The change in the levels of cfDNA/NETs across the NucleoCapture column at the end of each NucleoCapture treatment session.

SECONDARY OUTCOMES:
The amount of cfDNA/NETs in the circulating blood in patients after treatment with NucleoCapture compared to standard of care. | Within 6 hours from the baseline once 4.5 plasma volumes has been treated.
  The change in the levels of circulating cfDNA/NETS at the end of each NucleoCapture treatment session.
Change in organ in support | From date of randomisation to Day 5
  Change in organ support will be assessed by the combined change in Inotrope e.g. norepinephrine dose, lactate, urine output, Horowitz index and oxygenation index compared to standard of care
28-day survival | 28 days
  Survival up to 28 days
ICU length of stay | Up to 28 days.
  The length of stay in the ICU
Hospital length of stay | Up to 28 days
  The length of stay in up to hospital discharge

OTHER OUTCOMES:
Exploratory evaluation of the correlation between NucleoCapture treatment and levels of routine biomarkers. | At baseline, days 1 to 5, 7, 14 and 21.
  Routine organ function, haematology, coagulation and inflammation biomarkers will be measured.
Exploratory evaluation of the correlation between NucleoCapture treatment and levels of non-routine biomarkers. | At baseline, days 1 to 5, day 7 and day 14.
  Non-routine biomarkers of inflammation and coagulation will be measured.
Device handling and usability. | Day 1 to day 5.
  Usability and handling of the device will be assessed in the intervention arm using a questionnaire.
Patient reported outcome (PROMs) - PAN PROMISE acute pancreatitis symptom scale | Baseline, at discharge from the ICU up to day 28, and at 90 days post discharge from the ICU.
  Quantify the symptoms of acute pancreatitis via PROM.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szatmary, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No